CLINICAL TRIAL: NCT04762368
Title: Improving Vision in Adults With Macular Degeneration, Study 2: The Effect of Concurrent Perceptual Learning and Brain Stimulation
Brief Title: Learning Study: Improving Vision in Adults With Macular Degeneration
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Ben Thompson, Professor; Associate Director for Research, University of Waterloo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VSBrainStim2
Record Dates: First submitted 2021-02-13; First posted 2021-02-21 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-05

CONDITIONS: Macular Degeneration
Keywords: Macular Degeneration; Brain Stimulation; Psychophysics; Reading; tDCS; RSVP; Visual Acuity; Uncrowded Visual Acuity; Crowded Visual Acuity; Contrast Sensitivity
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Intervention Model Description: Group A: 6 training sessions with active brain stimulation and perceptual training Group B: 6 training sessions with sham brain stimulation and perceptual training
Who Masked: Participant, Investigator
Masking Description: The participant and the researcher will be blind to which group any given participant is assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active + Training (Active Comparator): Participants in this arm will be exposed to active stimulation for the first 25 minutes of a roughly hour - long perceptual training procedure in which participants must verbally read sentences presented at various speeds and sizes.
  Interventions: Device: Active anodal tDCS
- Sham + Training (Sham Comparator): Participants in this arm will be exposed to sham stimulation for the first 25 minutes of a roughly hour - long perceptual training procedure in which participants must verbally read sentences presented at various speeds and sizes.
  Interventions: Device: Sham anodal tDCS

INTERVENTIONS:
Device: Active anodal tDCS — a weak electric current is applied to the head through electrodes to affect the cortical excitability of the targeted cells in the brain.
  Arms: Active + Training
Device: Sham anodal tDCS — The tDCS machine will be used as in active stimulation, except the electrical current will not be applied.
  Arms: Sham + Training

SUMMARY:
The purpose of this study is to test whether a kind of brain stimulation called anodal transcranial direct current stimulation (a-tDCS) can be combined with perceptual learning to improve the ability of people with age-related macular degeneration (AMD) or juvenile macular degeneration (JMD) to read words presented to them on a computer screen better than if perceptual learning alone were used.

In addition, secondary measures of visual acuity will also be examined to determine whether brain stimulation can allow patients to resolve finer details of an image. The proposed treatment is the application of a-tDCS onto the participant's head, with brain stimulation aimed at Primary Visual Cortex toward the occipital pole, while patients undergo six separate sessions of training. The investigators will test the ability of participants to read words before the start of the training sessions (pre test) and after the completion of all training sessions (post test). This is a between-subjects design, and half of the participants will receive true stimulation, and the other half will receive sham stimulation. The difference between the pre and post tests when receiving active stimulation will be compared to the difference when receiving sham stimulation, because the sham stimulation is not expected to influence reading beyond a placebo. The aim of the study is to examine the potential of concurrent brain stimulation and perceptual learning as an effective treatment for macular degeneration that may be used in conjunction with more traditional eye-based interventions. The investigators hypothesize that the brain stimulation will enable higher performance in the reading task after and secondary measures after perceptual training due to an increase in the cortical excitability of the stimulated brain cells.

DETAILED DESCRIPTION:
This study will be carried out in Ontario, Canada (University of Waterloo) and Hong Kong (The Hong Kong Polytechnic University). There are two conditions: Active brain stimulation + perceptual training and sham/placebo brain stimulation + perceptual training. This study uses a between-subjects design, such that half of all participants will be placed in the active stimulation group and half will be placed in the sham group.

Participants will be recruited from university-affiliated clinics and local clinical practices. Following full informed consent, participants will complete baseline testing and clinical testing to confirm that they meet eligibility criteria including: a diagnosis of macular degeneration without any additional eye disease, impaired vision but with enough visual acuity that the computer monitor can still present readable word, and no contraindications for brain stimulation interventions. Eligible participants will then be randomized to either receiving the active stimulation during perceptual training or the placebo stimulation during perceptual training.

The primary outcome measure is verbal reading accuracy for sentences presented on a computer screen following a Rapid Serial Visual Presentation (RSVP) task in which a single word is presented on the screen at a time. Participants will freely observe the words and will indicate the words on the screen verbally. The secondary outcome measures are contrast sensitivity and crowded and uncrowded visual acuity as measured by Freiburg Visual Acuity & Contrast Test (FrACT) using the Landolt C stimulus. The "C"'s gap will be oriented randomly, and the participant will indicate the orientation of the stimulus. Crowded visual acuity will be assessed with Landolt C surrounded by a solid ring, while uncrowded visual acuity will be assessed with the Landolt C alone. The Test of contrast sensitivity will measure the amount of contrast required relative to the background to identify the orientation of the "C". The Hong Kong Polytechnic University has an additional set of secondary outcome measures of temporal and spatial visual span. Temporal visual span will be assessed using Chinese trigrams presented horizontally or vertically at the centre for a range of presentation times. Spatial visual span will be assessed using Chinese trigrams presented horizontally or vertically at different character positions for a fixed presentation time. Participants will be asked to recognize all three characters in a correct order.

The study consists of 9 sessions plus 1 additional session particularly for Hong Kong Polytechnic University

Session 0: This session only applies for The Hong Kong Polytechnic university, that horizontal and vertical temporal and spatial visual span will be collected.

Session 1: The first session will include the clinical evaluation. In addition, the pre tests of all outcome measures will be collected (RSVP performance, crowded and uncrowded visual acuity, contrast sensitivity).

Sessions 2-7: Brain stimulation sessions. Participants will undergo roughly 1 hour of perceptual training, performing the RSVP task. The first 25 minutes of this training will include either sham or active brain stimulation. A given participant will receive the same kind of stimulation for all 6 training sessions.

Session 8: No brain stimulation will occur. Post test outcome measures will be collected (RSVP performance, crowded and uncrowded visual acuity, contrast sensitivity, horizontal and vertical temporal and spatial visual span).

Session 9: 30 day follow up. 30 days after the final training session, participants will again perform the outcome measures without brain stimulation to determine the long term benefit of the perceptual training + brain stimulation.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of AMD (age 60+) or JMD (current age 18+).
2. Visual acuity (VA); between 6/9-6/96 in the better eye
3. Best-corrected near visual acuity of 4.0M at 40 cm or better in the better eye
4. Stable vision in previous 3 months (patient report)
5. Central vision loss

Exclusion Criteria:

1. Diagnosed dementia.
2. Not fluent in reading English (Waterloo) or Chinese characters (Hong Kong).
3. Any ocular surgery (including anti-vegF injections) within the duration of the study, except for: A. Chronic and continuous injections for at least 1 year. B. Injections stopped at least 2 months before participation. C. Injections in the untested eye
4. Ocular pathology other than JMD or AMD that can significantly reduce central vision. Example: mild cataract of grade 2 or below is acceptable
5. Severe hearing impairment.
6. Contraindications for brain stimulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-02-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Rapid Serial Visual Presentation (RSVP) Reading performance before and right after training. | The pre test and post test will take roughly 1 hour to complete, and they will be roughly 4-7 weeks apart.
  Behavioral Measure - Participants will verbally read words presented on a computer. A variety of speeds and sizes will be presented, so that an accurate measure of the maximum reading speed, and the smallest text size readable at the maximum reading speed can be calculated. The maximum reading speed and smallest text size will be measured before and after training. The outcome measures are the change in these reading measurements from pre test to post test.
Change in Rapid Serial Visual Presentation (RSVP) Reading performance 30 days after training | The test will take roughly 1 hour to complete, and they will be roughly 7-10 weeks apart.
  Behavioral Measure - Participants will verbally read words presented on a computer. A variety of speeds and sizes will be presented, so that an accurate measure of the maximum reading speed, and the smallest text size readable at the maximum reading speed can be calculated. The maximum reading speed and smallest text size will be measured before and after training. The outcome measures are the change in these reading measurements from pre test to the 30 day follow up.

SECONDARY OUTCOMES:
Change in Uncrowded Visual Acuity before and just after training | The pre test and post test will take roughly 5 minutes to complete, and they will be roughly 4-7 weeks apart.
  Visual acuity as measured by participants indicating the orientation of the gap present in a Landolt C stimulus using the freely available FrACT software https://michaelbach.de/fract/index.html . The outcome measure is the change in performance from pre test to the post test
Change in Uncrowded Visual Acuity before and 30 days after training | The pre test and post test will take roughly 5 minutes to complete, and they will be roughly 7 to 10 weeks apart.
  Visual acuity as measured by participants indicating the orientation of the gap present in a Landolt C stimulus using the freely available FrACT software https://michaelbach.de/fract/index.html . The outcome measure is the change in performance from pre test to the 30 day follow up.
Change in Crowded Visual Acuity before and just after training | The tests will take roughly 5 minutes to complete, and they will be roughly 4 - 7 weeks apart.
  Visual acuity as measured by participants indicating the orientation of the gap present in a Crowded (Ring) Landolt C stimulus using the freely available FrACT software https://michaelbach.de/fract/index.html . The outcome measure is the change in performance from pre test to post test.
Change in Crowded Visual Acuity before and 30 days after training | The tests will take roughly 5 minutes to complete, and they will be roughly 7 - 10 weeks apart.
  Visual acuity as measured by participants indicating the orientation of the gap present in a Crowded (Ring) Landolt C stimulus using the freely available FrACT software https://michaelbach.de/fract/index.html . The outcome measure is the change in performance from pre test to the 30 day follow up.
Change in Contrast Sensitivity before and just after training | The tests will take roughly 5 minutes to complete, and they will be roughly 4 - 7 weeks apart.
  Contrast sensitivity as measured by participants indicating the orientation of the gap present in a Landolt C stimulus using the freely available FrACT software https://michaelbach.de/fract/index.html . The outcome measure is the change in performance from pre test to the post test.
Change in Contrast Sensitivity before and 30 days after training | The tests will take roughly 5 minutes to complete, and they will be roughly 7-10 weeks apart.
  Contrast sensitivity as measured by participants indicating the orientation of the gap present in a Landolt C stimulus using the freely available FrACT software https://michaelbach.de/fract/index.html . The outcome measure is the change in performance from pre test to the 30 day follow up.
Change in Temporal Visual Span before and just after training | The test will take roughly 1.5 hours to complete, and they will be roughly 5-8 weeks apart
  Three unrelated Chinese characters will appear at the centre of a monitor for a range of exposure times. Participants will be asked to recognize all three characters in a correct order. Both horizontal and vertical presentation will be assessed. The outcome measures are the changes in time for recognizing the characters from pre test to the post test.
Change in Spatial Visual Span before and just after training | The test will take roughly 1.5 hours to complete, and they will be roughly 5-8 weeks apart.
  Three unrelated Chinese character will appear at different character positions for a fixed exposure time, while participants will be asked to keep fixation at the centre but recognize all three characters in a correct order. Both horizontal and vertical presentation will be assessed. The outcome measures are the changes in the size of the spatial visual span from pre test to the post.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Thompson, PhD, Principal Investigator — University of Waterloo
Locations (2):
- University of Waterloo, Waterloo, Ontario, Canada
- The Hong Kong Polytechnic University, Hung Hom, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
IDP that underlie results in a publication will be available after deidentification upon reasonable request to the research team.
Supporting Information: Analytic Code
Time Frame: IDP will be available upon a publication, and no more than 9 months after the publication.
Access Criteria: IDP will be shared to researchers who provide a methodologically sound proposal.

DOCUMENTS (2):
  • Study Protocol (2021-04-09): https://cdn.clinicaltrials.gov/large-docs/68/NCT04762368/Prot_002.pdf
  • Statistical Analysis Plan (2024-12-03): https://cdn.clinicaltrials.gov/large-docs/68/NCT04762368/SAP_003.pdf